CLINICAL TRIAL: NCT07332338
Title: Expanded Access Use of Human Umbilical Cord Blood (REGENECYTE) Infusion for Patients With Post-COVID Condition
Brief Title: Expanded Access Use of Human Umbilical Cord Blood (REGENECYTE) Infusion in Patients With Chronic Fatigue of Post-COVID Condition
Status: Temporarily not available | Type: Expanded Access
Sponsor: StemCyte, Inc. (Industry)
Responsible Party: Sponsor
Organization: StemCyte International, Ltd. (Industry)
Other Study IDs: SCUS001-EA1
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Post-COVID-19 Condition; Post-COVID Condition; Post-COVID Syndrome; Long COVID; Chronic Fatigue; Chronic Fatigue Symptoms; Fatigue Post Viral
Keywords: Long COVID; Post-COVID syndrome; Post-COVID condition; Umbilical cord blood; REGENECYTE; Post-COVID fatigue; Chronic fatigue symptoms; Fatigue post viral
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: REGENECYTE® — HPC, Cord Blood (Hematopoietic Progenitor Cell, Cord Blood)

SUMMARY:
REGENECYTE® (HPC, Cord Blood (Hematopoietic Progenitor Cell, Cord Blood)) for treatment in patients with post-COVID.

DETAILED DESCRIPTION:
A total of 30 subjects with post-COVID will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18
* With post-COVID condition
* Has had a recent (within 7 days) negative SARS-CoV-2 test (an approved PCR (polyermerase chain reaction) or antigen test)
* Not eligible for participation in any ongoing clinical trials of post-COVID condition with REGENECYTE
* Able to provide signed informed consent (by the subject or his/her legally authorized representative)
* Is willing and able to participate in all aspects of the study, including completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing a written informed consent

Exclusion Criteria:

* Neurological disorders prior to COVID-19 diagnosis
* With pre-existing terminal illness
* With known immune disease
* Is pregnant or breastfeeding
* Is currently participating in another investigational study or has been taking any other investigational product (IP) within the last 4 weeks before screening
* Has received any vaccination within 3 weeks prior to the first IP infusion or planning to receive vaccination during the treatment period
* Judged by the investigator to be not suitable for study participation, including but not limited to pre-existing chronic diseases
* Under the conditions that may increase risk of complications based on the medical judgment of the investigator and the parameters

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult